CLINICAL TRIAL: NCT04740567
Title: Early Cognitive Training and Rehabilitation to Improve Long-term Cognitive Outcomes in Older Hospitalized Adults With Delirium
Brief Title: Early Cognitive Intervention in Delirium
Acronym: ECID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Jin H. Han, Associate Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 192498
Record Dates: First submitted 2021-02-01; First posted 2021-02-05 (Actual); Results first posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Delirium; Cognitive Decline; Dementia
MeSH Terms: conditions — Delirium; Cognitive Dysfunction; Dementia | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Intervention (Experimental): During hospitalization, enrolled patients assigned to the intervention arm will undergo two 20-minute cognitive training sessions daily, 7 days a week. After the patient is discharged from the hospital, cognitive rehabilitation will be administered once a week for 12-weeks at their place of residence. Goal Management Training will be the foundation for cognitive rehabilitation.
  Interventions: Behavioral: Cognitive Training; Behavioral: Goal Management Training
- Usual Care (No Intervention): Enrolled patients will undergo usual care during hospitalization and post-hospital discharge.

INTERVENTIONS:
Behavioral: Cognitive Training — The cognitive training program regimen and its degree of difficulty will be tailored to the patient's current level of cognitive functioning and interests. Patients will be asked to work through progressively more challenging exercises pertaining to orientation, attention, problem-solving, and memory. These cognitive training exercises will be significantly difficult but when they can be completed easily (>85% mastery), their difficulty will be increased, and this process will be repeated as appropriate. They will also perform puzzles, games, or cognitive tasks related to their hobbies.
  Arms: Cognitive Intervention
Behavioral: Goal Management Training — Goal management training will (1) teach patients compensatory strategies such as "stop" techniques [e.g., to "stop and think" about consequences of a decision before making it]; (2) help them to take complex tasks and divide them into manageable subtasks to increase the likelihood of completing the task; and (3) enable them to learn to regain cognitive control when their behavior becomes incompatible with their intended goals. GMT is anchored in "sustained and vigilant attention theory" and it enables patients to actively attend to "higher order" goals critical to functioning. GMT is tailored to the individual needs of the patient. During the initial session, the Cognitive Intervention Specialist will meet with the subject and their family member or caregiver to identify these functional and cognitive deficiencies.
  Arms: Cognitive Intervention

SUMMARY:
This is a randomized control trial to determine if early cognitive training and rehabilitation improve 4-month cognition in hospitalized older (>=65 years old) delirious patients with and without Alzheimer's disease and related dementias. Enrolled patients will be randomized to receive cognitive intervention versus usual care at a 1:2 allocation ratio. Patients assigned to the cognitive intervention group will receive cognitive training daily during hospitalization and cognitive rehabilitation weekly for 12 weeks after hospital discharge. Patients will be evaluated for global cognition (primary outcome) and secondary outcomes at 4-months.

ELIGIBILITY:
Inclusion Criteria:

* 65 years or older
* Admitted through the ED
* Cognitive training can be initiated within 24 hours of ED presentation
* Delirious at enrollment

Exclusion Criteria:

* Comatose
* Not able to follow simple commands or non-verbal prior to the acute illness (end-stage pre-illness ADRD)
* Resides in a nursing home
* Prisoner
* Receiving hospice care
* Lives > 100 miles away from the enrolling sites
* Non-English speaking
* Previously enrolled
* Deaf or blind
* Intravenous drug, crack or cocaine, or methamphetamine use within the past one year, or any condition that, in the investigator's opinion, makes them an unreliable trial patient or unlikely to complete the trial.
* Psychotic disorder or suicidal gesture requiring hospitalization with the past one year
* Discharged from the ED

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 283 (Actual)
Dates: Start 2021-02-09 (Actual); Primary Completion 2024-11-14 (Actual); Study Completion 2024-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jin H Han, MD, MSc, Principal Investigator — Vanderbilt University Medical Center; James C Jackson, PsyD, Principal Investigator — Vanderbilt University Medical Center
Locations (2):
- United States (2):
  - Tennessee Valley Healthcare System - Nashville Veteran Affairs Hospital, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Deidentified data will be made available two years after publication. Supporting documents will be made available at the time of publication of the primary manuscript.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cognitive Intervention | Usual Care
Started (# randomized) | 97 | 186
Completed (# with primary outcome completed) | 50 | 102
Not Completed | 47 | 84
Not completed — Death | 31 | 43
Not completed — Lost to Follow-up | 2 | 11
Not completed — Patient declined to participate | 13 | 26
Not completed — Patient was physically incapable | 1 | 3
Not completed — Patient's spouse was had prolongued ICU stay | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive Intervention | Usual Care | Total
Number analyzed (Participants) | 97 | 186 | 283
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 97 | 186 | 283
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 76 [71 to 82] | 75 [70.3 to 82.0] | 75 [71 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 89 | 131
  Male | 55 | 97 | 152
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 14 | 27 | 41
  White | 81 | 154 | 235
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Global Cognition as Measured by the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS)
Description: A neuropsychological battery for global cognition which evaluates immediate and delayed memory, attention, visuospatial construction, and language. Scores range from 40 to 160, with higher scores indicating better cognition.
Time Frame: 4-months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Cognitive Intervention | Usual Care
Number analyzed (Participants) | 50 | 102
score on a scale | 67 [49 to 80] | 67 [52 to 83]

2. Secondary Outcome: Executive Function as Measured by the Components of the Delis-Kaplan Executive Function System (D-KEFS) Subscales
Description: The D-KEF's Proverbs, Color Word Interference, and Verbal Fluency Category Switching subscales will measure conceptual flexibility, inhibition, and monitoring, respecitvely, which encompasses the majority of executive function. The average of the three subscales will provide an executive function composite score. Scores range from 1 to 18 with higher values indicating better executive function
Time Frame: 4-months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Cognitive Intervention | Usual Care
Number analyzed (Participants) | 32 | 72
score on a scale | 5.5 [3 to 8] | 4.0 [0 to 11]

3. Secondary Outcome: Functional Status as Measured by Older American Resources and Services Activities of Daily Living Scale
Description: Characterizes seven basic and seven instrumental activities of daily living. Scores range from 0 to 28 with higher scores indicating better functional status.
Time Frame: 4-months
Population: Patient surrogates were able to complete this assessment which is why the total N is higher than the total number with completed outcomes.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Cognitive Intervention | Usual Care
Number analyzed (Participants) | 54 | 117
score on a scale | 9 [2 to 16] | 8 [3 to 13]

4. Secondary Outcome: Quality of Life as Measured by the EQ-5D-5L
Description: Characterizes quality of life and contains 5-dimensions ("5D") related to everyday living: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. It asks patients to rate their current global health status from 0 (worst health you can imagine) to 100 (best health you can imagine). Scores range from -0.573 to 1.000 with higher scores indicating better quality of life.
Time Frame: 4-months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Cognitive Intervention | Usual Care
Number analyzed (Participants) | 49 | 96
score on a scale | 0.352 [0.096 to 0.727] | 0.269 [0.096 to 0.465]

5. Secondary Outcome: Vital Status (Dead / Alive)
Description: Death within 4-months will be recorded
Time Frame: 4-months
Population: All patients who were randomized were included in the mortality outcome analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Cognitive Intervention | Usual Care
Number analyzed (Participants) | 97 | 186
Participants | 31 | 43

6. Secondary Outcome: Nursing Home Placement (Yes / no)
Description: Nursing home placement within 4-months will be recorded
Time Frame: 4-months
Population: All patients who were randomized included in the nursing home analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Cognitive Intervention | Usual Care
Number analyzed (Participants) | 97 | 186
Participants | 2 | 2

7. Secondary Outcome: Change in Montreal Cognitive Assessment
Description: Change in global cognition at 4-months compared to enrollment. The Montreal Cognitive Assessment assesses visuospatial, language, naming, memory, attention, abstraction, and orientation, and ranges from 0 to 30 (perfect cognition). It was collected at enrollment, during the delirium episode, and at 4 months.
Time Frame: 4-months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Cognitive Intervention | Usual Care
Number analyzed (Participants) | 40 | 85
score on a scale | 3.5 [0 to 6.5] | 4 [0 to 11]

ADVERSE EVENTS:
Time Frame: From enrollment to the 4-month follow-up
Arm/Group | Cognitive Intervention | Usual Care
All-Cause Mortality (participants affected / at risk) | 31/97 | 43/186
Serious Adverse Events (participants affected / at risk) | 0/97 | 0/186
Other Adverse Events (participants affected / at risk) | 0/97 | 0/186

LIMITATIONS AND CAVEATS:
Limited generalizability since our study was conducted at a quartnerary hospital in the South. Mortality was different between the intervention vs usual care group and overall attrition rate was high for both groups, which may have biased our estimates.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-02-04): https://cdn.clinicaltrials.gov/large-docs/67/NCT04740567/Prot_002.pdf
  • Statistical Analysis Plan (2024-11-14): https://cdn.clinicaltrials.gov/large-docs/67/NCT04740567/SAP_000.pdf
  • Informed Consent Form (2023-04-04): https://cdn.clinicaltrials.gov/large-docs/67/NCT04740567/ICF_003.pdf